CLINICAL TRIAL: NCT03140280
Title: A Pilot Study to Investigate the Hypomethylating Properties of Freeze-dried Black Raspberries (BRB) in Patients With Myelodysplastic Syndrome or Myelodysplastic Syndrome/Myeloproliferative Neoplasm (MDS/MPN)
Brief Title: Hypomethylating Properties of Freeze-dried Black Raspberries (BRB) in Patients With Myelodysplastic Syndrome or Myelodysplastic Syndrome/Myeloproliferative Neoplasm (MDS/MPN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ehab L Atallah (Other)
Responsible Party: Sponsor-Investigator, Ehab L Atallah, Professor, Department of Medicine, Division of Hematology/Oncology, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO28985
Record Dates: First submitted 2017-02-23; First posted 2017-05-04 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: Black raspberries; MDS; Myelodysplastic Syndromes; hypomethylating effects; chemopreventive agent; BRB; pharmacokinetics
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dietary Intervention (Experimental): Freeze-dried black raspberry powder administration.
  Interventions: Drug: Freeze-Dried Black Raspberry Powder

INTERVENTIONS:
Drug: Freeze-Dried Black Raspberry Powder — 25 gm (2x/day) of freeze-dried black raspberry powder taken orally in 8 ounces of water for 12 weeks. If the patient is tolerating BRBs well and is benefiting from therapy, he or she will continue treatment for a total maximum of 48 weeks.

SUMMARY:
This is a phase II, single-group pilot study to evaluate efficacy and methylation. This study's overarching aim is to evaluate the systemic effects of black raspberries in patients with myelodysplastic syndrome or myelodysplastic syndrome/myeloproliferative neoplasm. Twenty-one patients with MDS will be treated with 25 gm (2x/day) of BRB powder taken orally.

DETAILED DESCRIPTION:
STUDY RATIONALE:

Hypomethylating agents (HMAs) such as azacitidine and decitabine are FDA approved therapies for MDS patients. Approximately 50% of patients respond to HMAs. In addition, HMAs have improved survival and quality of life of patients with MDS when compared with other therapies.

Preclinical research shows black raspberries (BRBs) have hypomethylating effects in the colon, blood, spleen, and bone marrow of mice treated with BRBs. The aim of this study is to evaluate the hypomethylating properties of BRBs in patients with MDS or MDS/MPN for three cycles (one cycle = 28 days) of BRB supplementation.

PRIMARY OBJECTIVE:

To evaluate the potential hypomethylating effects of freeze-dried black raspberries (BRBs) in the peripheral blood of patients with myelodysplastic syndrome or myelodysplastic syndrome/myeloproliferative neoplasm (MDS/MPN) after three cycles of BRB administration.

SECONDARY OBJECTIVE:

1. To evaluate the toxicity of BRBs in patients with MDS or MDS/MPN.
2. To evaluate the hematological response according to modified International Working Group (IWG) criteria (Appendix 2) in patients with MDS or MDS/MPN regardless of the initial blood count.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a confirmed diagnosis of myelodysplastic syndrome or myelodysplastic syndrome/myeloproliferative neoplasm (MDS/MPN) proven by bone marrow biopsy/aspirate.
2. Patients with cytopenias (blood cell counts lower than the institutional lower limit of normal within the eight weeks prior to the study) who are receiving or received:

   * red blood cell transfusions
   * observation
   * platelet transfusions
   * erythropoietin
   * granulocyte colony-stimulating factors
   * granulocyte-macrophage colony-stimulating factors
   * hydrea
3. Age >18 years.
4. Predicted life expectancy of at least 12 weeks.
5. Patients should be expected to stay on the same therapy for the period of the study.
6. Patients who do not have an indication for and/or are unable to tolerate a hypomethylating agent are eligible for the study.
7. Reproductive requirements:

   Female patients must meet one of the following:
   * Postmenopausal for at least one year before the screening visit, or
   * Surgically sterile, or
   * If women are of childbearing potential, agree to practice two effective methods of contraception from the time of signing of the informed consent form through 30 days after the last dose of study drug, AND
   * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, or
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable contraception methods.)

   Male patients, even if surgically sterilized (i.e., status postvasectomy), must agree to one of the following:
   * Practice effective barrier contraception during the entire study treatment period and through 30 days after the last study drug dose, OR
   * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)
8. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

A potential subject who meets any of the following exclusion criteria is ineligible to participate in the study.

1. Previously received hypomethylating agents.
2. Allergy to black raspberries.
3. Inability to swallow oral medication.
4. Inability or unwillingness to comply with the BRB administration requirements.
5. Uncontrolled intercurrent illness, including, but not limited to, symptomatic congestive heart failure, or psychiatric illness/social situations, that, in the treating investigator's discretion, would limit compliance with study requirements.
6. Active infection not well controlled by antibacterial or antiviral therapy.
7. Pregnant or lactating women.
8. Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Atallah, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dietary Intervention
Started | 23
Completed | 18
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | Dietary Intervention
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Grade 3 or Higher Serious Adverse Events.
Description: Adverse events assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0; patients will be evaluated every four weeks for toxicity.
Time Frame: Up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dietary Intervention
Number analyzed (Participants) | 18
Participants | 3

2. Secondary Outcome: The Number of Subjects Showing a Response.
Description: The subject's best clinical response will be assessed based on the modified International Working Group response criteria while receiving BRBs.
Time Frame: Up to 52 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dietary Intervention
Number analyzed (Participants) | 18
Participants | 0

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: This measure reports serious adverse events regardless of grade.
Arm/Group | Dietary Intervention
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 4/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dietary Intervention (N=18)
Syncope (Nervous system disorders) | 1 (1)
Allergic Reaction (Immune system disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Death not otherwise specified (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dietary Intervention (N=18)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Alanine transaminase increased (Investigations) | 2 (2)
alkaline phosphatase increased (Investigations) | 3 (4)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (6)
Aspartate transferase increase (Investigations) | 2 (3)
Bloating (Gastrointestinal disorders) | 3 (3)
Blood bilirubin increase (Investigations) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 4 (5)
Chills (General disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Fatigue (General disorders) | 5 (6)
Flatulence (Gastrointestinal disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (2)
Gastrointestional disorders other, specify (Gastrointestinal disorders) | 1 (1) — Thrush
Headache (Nervous system disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hepatobiliary disorders, specify (Hepatobiliary disorders) | 1 (1) — Increased lactate dehydrogenase
Hyperglycemia (Metabolism and nutrition disorders) | 6 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
Hypermagnasemia (Metabolism and nutrition disorders) | 1 (2)
Hypertension (Vascular disorders) | 4 (5)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestations, other, specify (Infections and infestations) | 1 (1) — Influenza
Injury, poisoning and procedural complications, other, specify (Injury, poisoning and procedural complications) | 1 (1) — Splenic rupture
Injury, poisoning and procedural complications, other, specify (Injury, poisoning and procedural complications) | 1 (1) — Ecchymosis
Insomnia (Psychiatric disorders) | 1 (1)
Investigations, other, specify (Investigations) | 2 (2) — Decreased creatinine
Lymphedema (Vascular disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (12)
Metabolism and nutrition disorders, others, specify (Metabolism and nutrition disorders) | 1 (1) — Decreased total protein
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps), other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — breast cancer
Neutrophil count decreased (Investigations) | 9 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 1 (1)
Platlet count decrease (Investigations) | 5 (13)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders, other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Rhinorrhea
Sinus bradycardia (Cardiac disorders) | 1 (1)
Skin and subcutaneous tissue disorders, other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Plantar wart
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
White blood cell count decreased (Investigations) | 7 (17)
Edema limbs (General disorders) | 2 (3)
Intra-abdominal hemmorrhage (Gastrointestinal disorders) | 1 (1)
Localized edema (General disorders) | 2 (3)
Non-cardiac chest pain (General disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-12-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT03140280/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/80/NCT03140280/ICF_001.pdf